CLINICAL TRIAL: NCT06551168
Title: The Cardiovascular, Hematological, and Performance Response to Heat Acclimation in Healthy Trained Females
Brief Title: Heat Acclimation in Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Western University (Other)
Responsible Party: Principal Investigator, Anita Cote, Associate Professor, Trinity Western University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22G18
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Heat Exposure; Blood Volume; Cardiac Output
Keywords: basic science
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The experimental group will undergo heat acclimation The control group will not undergo heat acclimation. The control group will undergo heart rate matched exercise of the same quantity but in a cool environment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heat Acclimation (Experimental): Participants in this arm will undergo heat acclimation sessions
  Interventions: Other: Heat exposure
- Control (Active Comparator): Participants in this arm will undergo heart rate matched training volume
  Interventions: Other: Control group

INTERVENTIONS:
Other: Heat exposure — Participants will exercise at home while wearing a clothing ensemble over 19 one hour sessions. They will use validated perceptual scales to guide their effort and thermal sensation.
  Arms: Heat Acclimation
Other: Control group — Participants will exercise at home over 19 one hour sessions. They will use heart rate to guide their effort. The exercise will take place in cool conditions
  Arms: Control

SUMMARY:
Heat acclimation is when you repeatedly exposure yourself to heat so that your body adapts and better tolerates heat.

This project will determine if completing a heat acclimation maintenance period after heat acclimation is more beneficial than heat acclimating alone for exercise performance in the heat. To determine this, participants will exercise in the heat before heat acclimation, after heat acclimation, and after heat acclimation maintenance. Researchers will assess the heart's pumping capacity, blood volume, body temperature, and exercise performance to determine which approach is more effective.

DETAILED DESCRIPTION:
Purpose and Hypothesis: Global warming combined with increased frequency of heat waves exposes those who are working, exercising, or competing outdoors to considerable thermal strain. Excessive heat stress decreases exercise performance and can lead to heat illnesses. Deliberate serial exposure to natural (acclimatization) or artificial (acclimation) heat (HA) is the most efficacious method to defend homeostasis at rest and during exercise in hot environments. Our project will determine if three weeks of heat acclimation maintenance (HAM) further potentiates exercise performance in the heat than exercise performance measured after 10 days of HA in females.

Justification: Female participation in arduous occupations and professional sport is increasing. Presently a paucity of data regarding the female response to heat acclimation exist. Findings from this study will help females undertake effective and efficient strategies to mitigate thermal strain.

Research design: This is an experimental trial with a treatment and a control group. VO2max, plasma volume (PV), core temperature, and cardiac output will be measured pre-, mid-, and post-intervention. Participants will complete 10 sessions of HA over two weeks. Participants will then undergo three weeks of HAM with three heat sessions per week. A heat performance test will be completed pre-, mid-, and post-intervention to examine performance changes. A control group will complete the same test schedule but will not perform any HA or HAM.

Statistical analysis: Sample size will be 8 females in the experimental and 6 females in the control group. Data will be analyzed for normality using the Shapiro-Wilk test. Descriptive statistics will be presented as the mean and standard deviation. Statistical significance will be determined at P <0.05. A two-way repeated measure ANOVA will be used to measure differences between groups and hemodynamic, cardiovascular and performance variable differences pre- and post-HA, and pre- post-HAM. If significant effects are present, these will be followed by a post-hoc Tukey's test. Pearson's r correlations (two-tailed) will be conducted between VO2max, and intravascular volumes and heat performance test outcome.

ELIGIBILITY:
Inclusion Criteria:

* Familiar with the sport of cycling and own a bicycle and smart trainer (or a trainer and a power meter).
* Endurance athlete or currently engaging in endurance exercise
* Maximal oxygen consumption (VO2max) greater than 40 ml/kg/min
* Between the ages of 18 and 55
* Able to speak, read, and write in English

Exclusion Criteria:

* Unable to exercise
* Previous or current heat intolerance
* Pregnant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Performance | 2 weeks and 5 weeks
  Participants will complete a timetrial on a cycle ergometer in a heat chamber. Faster times following HA or HAM will be considered a marker of performance

SECONDARY OUTCOMES:
Intravascular volumes | 2 weeks and 5 weeks
  Expanded plasma volume or increased hemoglobin mass will be considered a positive response to heat acclimation

CONTACTS AND LOCATIONS:
Overall Officials: Anita T Coté, PhD, Principal Investigator — Trinity Western University
Locations (1):
- Trinity Western Unversity, Langley, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided